CLINICAL TRIAL: NCT03361046
Title: Evaluation of Clinical Outcomes of Transcatheter Aortic Valve-in-Valve Implantation in Polish Population - Observational Multicenter Registry
Brief Title: Polish Transcatheter Aortic Valve-in-Valve Implantation (ViV-TAVI) Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: WUM-VIV
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Insufficiency; Ventricular Outflow Obstruction, Left
Keywords: TAVI; valve-in-valve; aortic stenosis
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency; Ventricular Outflow Obstruction, Left

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Transcatheter Aortic Valve-in-Valve Implantation Cohort
  Interventions: Device: Transcatheter Aortic Valve-in-Valve Implantation (ViV-TAVI)

INTERVENTIONS:
Device: Transcatheter Aortic Valve-in-Valve Implantation (ViV-TAVI) — Patients with failed aortic valve bioprostheses qualified for TAVI due to coexisting illnesses
  Other Names: Transcatheter Aortic Valve-in-Valve Replacement (ViV-TAVR)

SUMMARY:
In the past years a substantial shift away from mechanical heart valves occurred and bioprosthetic heart valves claimed majority of market shares irrespective of patients' age.This indicates that population with failed surgical bioprostheses requiring ViV-TAVI will grow significantly and therefore, meticulous prospective data collection is necessary for future analyses in order to better understand potential limitations of this procedure.

DETAILED DESCRIPTION:
The study is a prospective multicenter evaluation of transcatheter aortic valve-in-valve implantations in Polish health centers.

Duration of this study is expected to be 6 years to ensure that all of the enrolled patients will complete at least 2 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Failing surgically implanted aortic bioprosthetic valve (stented/stentless/homograft) demonstrating ≥ moderate stenosis and/or ≥ moderate insufficiency
* Qualification for TAVI by decision of the local Heart Team
* Patient provided written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients meeting inclusion criteria will prospectively included in the study. Patients meeting inclusion criteria before the set-up of registry will be included retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
VARC (Valve Academic Research Consortium-2) defined "Clinical Efficacy" composite endpoint | From 30 days post procedure to completion of at least 2 years of follow up
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Requiring hospitalizations for valve-related symptoms or worsening congestive heart failure
  * NYHA (New York Heart Association) class III or IV functional classification of heart failure
  * Valve-related dysfunction (mean aortic valve gradient ≥20 mmHg, Effective Orifice Area (EOA) ≤0.9-1.1 cm2(c) and/or Doppler Velocity Integral (DVI) <0. 35 m/s, AND/OR moderate or severe prosthetic valve regurgitation

SECONDARY OUTCOMES:
VARC defined 'Device success' composite endpoint | 30 days
  * Absence of procedural mortality AND
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location AND
  * Intended performance of the prosthetic heart valve (no prosthesis - patient mismatch and mean aortic valve gradient ,20 mmHg or peak velocity ,3 m/s, AND no moderate or severe prosthetic valve regurgitation)
VARC defined "Early Safety" composite endpoint | 30 days
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Life-threatening bleeding
  * Acute kidney injury-Stage 2 or 3 (including renal replacement therapy)
  * Coronary artery obstruction requiring intervention
  * Major vascular complication
  * Valve-related dysfunction requiring repeat procedure (Balloon Aortic Valvuloplasty (BAV), Trans Catheter Aortic Valve Implant (TAVI), or Surgical Aortic Valve Replacement (SAVR))
VARC defined "Time-related valve safety" composite endpoint | From device implant to completion of at least 2 years of follow up
  * Structural valve deterioration
  * Valve-related dysfunction (mean aortic valve gradient ≥20 mmHg, EOA ≤0.9-1.1 cm2cand/or DVI <0.35 m/s, AND/OR moderate or severe prosthetic valve regurgitation)
  * Requiring repeat procedure (TAVI or SAVR)
  * Prosthetic valve endocarditis
  * Prosthetic valve thrombosis
  * Thrombo-embolic events (e.g. stroke)
  * VARC bleeding, unless clearly unrelated to valve therapy (e.g. trauma)

CONTACTS AND LOCATIONS:
Overall Officials: Zenon Huczek, MD, PhD, Principal Investigator — Medical University of Warsaw; Wojciech Wojakowski, MD, PhD, Principal Investigator — Medical University of Silesia
Locations (12):
- Poland (12):
  - Medical University of Bialystok, Bialystok
  - Polish-American Heart Clinic, Bielsko-Biala
  - Medical University of Gdansk, Gdansk
  - Medical University of Silesia, Katowice
  - Jagiellonian University Medical College, Krakow
  - Medical University of Lodz, Lodz
  - Poznan University of Medical Sciences, Poznan
  - District Hospital 2, Rzeszów
  - Institute of Cardiology, Warsaw
  - Medical University of Warsaw, Warsaw
  - Wroclaw Medical University, Wroclaw
  - Silesian Center for Heart Diseases, Zabrze

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kappetein AP, Head SJ, Genereux P, Piazza N, van Mieghem NM, Blackstone EH, Brott TG, Cohen DJ, Cutlip DE, van Es GA, Hahn RT, Kirtane AJ, Krucoff MW, Kodali S, Mack MJ, Mehran R, Rodes-Cabau J, Vranckx P, Webb JG, Windecker S, Serruys PW, Leon MB; Valve Academic Research Consortium (VARC)-2. Updated standardized endpoint definitions for transcatheter aortic valve implantation: the Valve Academic Research Consortium-2 consensus document (VARC-2). Eur J Cardiothorac Surg. 2012 Nov;42(5):S45-60. doi: 10.1093/ejcts/ezs533. Epub 2012 Oct 1. PMID 23026738
- [Background] McElhinney DB, Cabalka AK, Aboulhosn JA, Eicken A, Boudjemline Y, Schubert S, Himbert D, Asnes JD, Salizzoni S, Bocks ML, Cheatham JP, Momenah TS, Kim DW, Schranz D, Meadows J, Thomson JD, Goldstein BH, Crittendon I 3rd, Fagan TE, Webb JG, Horlick E, Delaney JW, Jones TK, Shahanavaz S, Moretti C, Hainstock MR, Kenny DP, Berger F, Rihal CS, Dvir D; Valve-in-Valve International Database (VIVID) Registry. Transcatheter Tricuspid Valve-in-Valve Implantation for the Treatment of Dysfunctional Surgical Bioprosthetic Valves: An International, Multicenter Registry Study. Circulation. 2016 Apr 19;133(16):1582-93. doi: 10.1161/CIRCULATIONAHA.115.019353. Epub 2016 Mar 18. PMID 26994123
- [Result] Huczek Z, Grodecki K, Scislo P, Wilczek K, Jagielak D, Fil W, Kubler P, Olszowka P, Dabrowski M, Frank M, Grygier M, Kidawa M, Wilimski R, Zelazowska K, Witkowski A, Kochman J, Zembala M, Opolski G, Dvir D, Wojakowski W. Transcatheter aortic valve-in-valve implantation in failed stentless bioprostheses. J Interv Cardiol. 2018 Dec;31(6):861-869. doi: 10.1111/joic.12540. Epub 2018 Jul 15. PMID 30009390
- [Result] Scislo P, Grodecki K, Binczak D, Kochman J, Wilimski R, Huczek Z. Valve-in-valve treatment of dysfunctional aortic bioprostheses - single-centre experience. Postepy Kardiol Interwencyjnej. 2018;14(4):425-428. doi: 10.5114/aic.2018.79872. Epub 2018 Dec 11. No abstract available. PMID 30603033
- [Derived] Jonik S, Mazurek M, Rymuza B, Jankowski J, Dabrowski M, Wolny R, Chodor P, Wilczek K, Fil W, Milewski K, Protasiewicz M, Sciborski K, Kaplon-Cieslicka A, Skrobucha A, Hawranek M, Scislo P, Wilimski R, Kochman J, Grabowski M, Grygier M, Witkowski A, Huczek Z. Redo-Transcatheter Aortic Valve Implantation (Redo-TAVI)-Pilot Study from Multicentre Nationwide Registry. J Clin Med. 2025 Nov 14;14(22):8078. doi: 10.3390/jcm14228078. PMID 41303113